CLINICAL TRIAL: NCT01103219
Title: Nutrition, Growth and Development Among Very Preterm Infants
Acronym: PRENU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: A planned interim-analysis revealed increased number of infections in the intervention arm.
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Per Ole Iversen, MD, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRENU-1
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Low Birth Weight Infant
Keywords: VLBW; nutrition; vitamin A; long-chain unsaturated fatty acids; growth; cognitive functions; Very low birth weight infants (birth weight below 1,500 grams).
MeSH Terms: interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Participants in this group will receive nutrition from birth and during the hospital stay until discharge according to the routines of the participating institutions.
  Interventions: Dietary Supplement: Nutrition
- Intervention (Active Comparator): The participants in this group will receive increased supply of energy, protein, vitamin A, docosahexaenoic acid, and arachidonic acid from birth and during the hospital stay until discharge.
  Interventions: Dietary Supplement: Nutrition

INTERVENTIONS:
Dietary Supplement: Nutrition — The control (placebo) group will be fed according to the routines of the participating institutions. The intervention (active) group will receive increased supply of energy, protein, vitamin A and long-chain unsaturated fatty acids.

SUMMARY:
The main purpose of this study is to evaluate the effect of increased supply of energy, protein, vitamin A and the long chain polyunsaturated fatty acids docosahexaenoic acid and arachidonic acid on growth, brain maturation and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight below 1,500 grams
* Written consent to participate from the parents

Exclusion Criteria:

* Congenital malformations
* Clinical syndromes known to affect growth and development
* Critical illness and short life expectancy
* If participants refuse to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-08; Primary Completion 2012-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Reduction in discharge rate of small-for-gestational age very low birth weight infants | 6 months corrected age
  The primary endpoint is to reduce the discharge rate of very low birth weight infants that are small-for-gestational age, from 60 to 40%.

SECONDARY OUTCOMES:
Evaluation of brain function and growth of infant | 6 months corrected age
  Secondary endpoints will include:
  1. Assessment of brain maturation using MRI.
  2. Cognitive measurements.
  3. Anthropometric measures and biomarkers to assess body growth and development.
  4. Morbidity- (e.g. ROP, BPD, PVL, NEC) and mortality rates.

CONTACTS AND LOCATIONS:
Overall Officials: Per O Iversen, MD, Principal Investigator — University of Oslo
Locations (3):
- Norway (3):
  - Akershus University Hospital, Nordbyhagen
  - Oslo University Hospital, Rikshospitalet, Oslo
  - Oslo University Hospital, Ullevaal, Oslo

REFERENCES:
- [Background] Westerberg AC, Henriksen C, Ellingvag A, Veierod MB, Juliusson PB, Nakstad B, Aurvag AK, Ronnestad A, Gronn M, Iversen PO, Drevon CA. First year growth among very low birth weight infants. Acta Paediatr. 2010 Apr;99(4):556-62. doi: 10.1111/j.1651-2227.2009.01667.x. Epub 2010 Jan 20. PMID 20096031
- [Background] Henriksen C, Westerberg AC, Ronnestad A, Nakstad B, Veierod MB, Drevon CA, Iversen PO. Growth and nutrient intake among very-low-birth-weight infants fed fortified human milk during hospitalisation. Br J Nutr. 2009 Oct;102(8):1179-86. doi: 10.1017/S0007114509371755. Epub 2009 May 18. PMID 19445820
- [Background] Henriksen C, Haugholt K, Lindgren M, Aurvag AK, Ronnestad A, Gronn M, Solberg R, Moen A, Nakstad B, Berge RK, Smith L, Iversen PO, Drevon CA. Improved cognitive development among preterm infants attributable to early supplementation of human milk with docosahexaenoic acid and arachidonic acid. Pediatrics. 2008 Jun;121(6):1137-45. doi: 10.1542/peds.2007-1511. PMID 18519483
- [Background] Aurvag AK, Henriksen C, Drevon CA, Iversen PO, Nakstad B. Improved vitamin A supplementation regimen for breastfed very low birth weight infants. Acta Paediatr. 2007 Sep;96(9):1296-302. doi: 10.1111/j.1651-2227.2007.00445.x. PMID 17718782
- [Background] Henriksen C, Helland IB, Ronnestad A, Gronn M, Iversen PO, Drevon CA. Fat-soluble vitamins in breast-fed preterm and term infants. Eur J Clin Nutr. 2006 Jun;60(6):756-62. doi: 10.1038/sj.ejcn.1602379. Epub 2006 Feb 1. PMID 16452918
- [Background] Westerberg AC, Schei R, Henriksen C, Smith L, Veierod MB, Drevon CA, Iversen PO. Attention among very low birth weight infants following early supplementation with docosahexaenoic and arachidonic acid. Acta Paediatr. 2011 Jan;100(1):47-52. doi: 10.1111/j.1651-2227.2010.01946.x. PMID 20624152
- [Derived] Amissah EA, Brown J, Harding JE. Protein supplementation of human milk for promoting growth in preterm infants. Cochrane Database Syst Rev. 2020 Sep 23;9(9):CD000433. doi: 10.1002/14651858.CD000433.pub3. PMID 32964431
- [Derived] Strommen K, Haag A, Moltu SJ, Veierod MB, Blakstad EW, Nakstad B, Almaas AN, Braekke K, Ronnestad AE, Daniel H, Drevon CA, Iversen PO. Enhanced nutrient supply to very low birth weight infants is associated with higher blood amino acid concentrations and improved growth. Clin Nutr ESPEN. 2017 Apr;18:16-22. doi: 10.1016/j.clnesp.2017.01.003. Epub 2017 Feb 13. PMID 29132733
- [Derived] Blakstad EW, Moltu SJ, Nakstad B, Veierod MB, Strommen K, Juliusson PB, Almaas AN, Ronnestad AE, Braekke K, Drevon CA, Iversen PO. Enhanced nutrition improves growth and increases blood adiponectin concentrations in very low birth weight infants. Food Nutr Res. 2016 Dec 1;60:33171. doi: 10.3402/fnr.v60.33171. eCollection 2016. PMID 27914187
- [Derived] Strommen K, Lyche JL, Blakstad EW, Moltu SJ, Veierod MB, Almaas AN, Sakhi AK, Thomsen C, Nakstad B, Braekke K, Ronnestad AE, Drevon CA, Iversen PO. Increased levels of phthalates in very low birth weight infants with septicemia and bronchopulmonary dysplasia. Environ Int. 2016 Apr-May;89-90:228-34. doi: 10.1016/j.envint.2016.01.024. Epub 2016 Feb 26. PMID 26922148
- [Derived] Moltu SJ, Strommen K, Blakstad EW, Almaas AN, Westerberg AC, Braekke K, Ronnestad A, Nakstad B, Berg JP, Veierod MB, Haaland K, Iversen PO, Drevon CA. Enhanced feeding in very-low-birth-weight infants may cause electrolyte disturbances and septicemia--a randomized, controlled trial. Clin Nutr. 2013 Apr;32(2):207-12. doi: 10.1016/j.clnu.2012.09.004. Epub 2012 Sep 21. PMID 23043722